CLINICAL TRIAL: NCT03054402
Title: Randomized, Placebo-controlled, Double-blind Study to Investigate the Safety, Tolerability, Pharmacokinetics and to Explore Pharmacodynamics of Increasing Single Oral Doses of BAY1834845 Including Relative Bioavailability of a Liquid Versus a Solid Dosage in Healthy Male Volunteers
Brief Title: First in Human Study to Investigate the Safety, Tolerability, Pharmacokinetics and to Explore Pharmacodynamics of BAY1834845
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18384; 2016-002668-15 (EudraCT Number)
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Inflammatory Disease
MeSH Terms: conditions — Pelvic Inflammatory Disease | interventions — zabedosertib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation/BAY1834845 (Experimental): Subjects will receive a single dose of BAY1834845 in the morning of the PK profile day
  Interventions: Drug: BAY1834845
- Placebo (Placebo Comparator): Subjects will receive a single dose of placebo in the morning of the PK profile day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1834845 — Escalating doses of BAY1834845 including comparison of solution and tablet in one dose group
  Arms: Dose escalation/BAY1834845
Drug: Placebo — Single dose of placebo
  Arms: Placebo

SUMMARY:
This study is a first in human study that will investigate the safety, tolerability and pharmacokinetics and explore the pharmacodynamics of ascending single doses of BAY1834845 using a placebo controlled, randomized, single center design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 50 years (inclusive) at the first screening visit
* Body mass index (BMI) : 18.5 ≤ BMI ≤ 30 kg/m²

Exclusion Criteria:

* Clinically relevant findings in the physical examination
* Relevant diseases within the last 4 weeks prior to the first study drug administration
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Use of systemic or topical medicines or substances which oppose the study objectives or which might influence them within 4 weeks before first study drug administration

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events (TEAEs) | Up to 25 days after last drug administration
  AEs are considered to be treatment-emergent if they have started or worsened after first application of study medication up to 30 days after end of treatment with study medication.
Severity of treatment-emergent adverse events | Up to 25 days after last drug administration
  The intensity of an AE is classified according to the following categories:
  * Mild
  * Moderate
  * Severe
Area under the plasma concentration vs. time curve (AUC) | Baseline to up to 14 days post drug administration
  AUC from zero to infinity after single dose if possible or from time 0 to the last data point above lower limit of quantification (AUC (0-tlast)
Maximum drug concentration in plasma after single dose administration (Cmax) | Baseline to up to 14 days post drug administration
  Maximum drug concentration in plasma in mg/L after single dose administration of BAY1834845

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

REFERENCES:
- [Derived] Feldmuller M, Jodl SJ, Ploeger B, Wagenfeld A, Wiesinger H, Zollmann FS, Klein S, Zhang R, Rohde B, Hochel J. Zabedosertib, a novel interleukin-1 receptor-associated kinase-4 inhibitor, shows a favorable pharmacokinetic and safety profile across multiple phase 1 studies. Front Pharmacol. 2025 May 30;16:1521505. doi: 10.3389/fphar.2025.1521505. eCollection 2025. PMID 40520205